CLINICAL TRIAL: NCT04054479
Title: The Effect of Penehyclidine on Postoperative Nausea and Vomiting After Strabismus Surgery
Brief Title: Penehyclidine for PONV Prophylaxis After Strabismus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-SR-238
Record Dates: First submitted 2019-08-11; First posted 2019-08-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: PONV
Keywords: Penehyclidine; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — penehyclidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penehyclidine (Experimental): Patients in this arm will receive penehyclidine after anesthesia intubation.
  Interventions: Drug: Penehyclidine
- Normal Saline (Placebo Comparator): Patients in this arm will receive normal saline after anesthesia intubation.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Penehyclidine — Patients receive penehyclidine 10μg/kg(up to 0.5mg, diluted with normal saline to 0.1mg/ml) after anesthesia intubation.
  Arms: Penehyclidine
Drug: normal saline — Patients receive 0.1ml/kg normal saline(up to 5ml) after anesthesia intubation.
  Arms: Normal Saline

SUMMARY:
Patients scheduled for elective strabismus surgery under general anesthesia in the First Affiliated Hospital of Nanjing Medical University will be included in this study.

Patients 1)ASA I or II, 2)aged 3-65 years, 3)scheduled for elective strabismus surgery under general anesthesia, will be included in the study. Patients 1)had prior PONV, 2)severe motion sickness, 3)a history of ophthalmic surgery, 4)had received drugs known to have antiemetic effects, will be excluded from the study.

The primary aim is to evaluate the prophylaxis effect of penehyclidine(a novel long acting selective anticholinergic agent developed in China) on postoperative nausea and vomiting after strabismus surgery. Secondary outcomes include the effect of PONV risk factors and surgical technique on PONV rank score, occurance of oculocardiac reflex, time to extubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Aged 3-65 years
* Scheduled for elective strabismus surgery under general anesthesia

Exclusion Criteria:

* Had prior PONV
* Severe motion sickness
* A history of ophthalmic surgery
* Had received drugs known to have antiemetic effects in 24h before surgery

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV | From extubation to 48 hours after surgery
  Occurance of postoperative nausea and vomiting after strabismus surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhengnian Ding, M.D., Study Chair — The First Affiliated Hospital with Nanjing Medical University; Xiaofei Cao, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Ting Lu, M.M., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Jiacheng Sun, M.M., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun J, Cao X, Lu T, Li N, Min X, Ding Z. Penehyclidine mitigates postoperative nausea and vomiting and intraoperative oculocardiac reflex in patients undergoing strabismus surgery: a prospective, randomized, double-blind comparison. BMC Anesthesiol. 2021 Feb 13;21(1):49. doi: 10.1186/s12871-021-01266-0. PMID 33581727